CLINICAL TRIAL: NCT02454322
Title: The Effect of Magnesium on Maternal Mood, Cognitive Function, and Birth Experience
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Emily Miller, Assistant Professor in Obstetrics and Gynecology-Maternal Fetal Medicine and Psychiatry and Behavioral Sciences, Northwestern University
Other Study IDs: IRB #200388
Record Dates: First submitted 2015-05-15; First posted 2015-05-27 (Estimated); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Depression, Postpartum
MeSH Terms: conditions — Depression, Postpartum | interventions — Magnesium Sulfate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cerebrospinal fluid and peripheral serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Magnesium: Hypertensive Disorder of Pregnancy (gestational hypertension or preeclampsia) Treated with Magnesium Sulfate
  Interventions: Drug: Magnesium Sulfate
- No Magnesium: Hypertensive Disorder of Pregnancy (gestational hypertension or preeclampsia) Not Treated with Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — Standard of care Magnesium Sulfate given to women with a diagnosis of a hypertensive disorder of pregnancy.
  Groups: Magnesium

SUMMARY:
Magnesium is sometimes used to prevent seizures in the setting of hypertensive disorders of pregnancy. The primary aim of this study is to determine if women who receive magnesium are less likely to experience postpartum depression. Other aims include examining the relationship between receiving magnesium and cognitive function and birth experience.

DETAILED DESCRIPTION:
This prospective observational study of women with hypertensive disorders of pregnancy (gestational hypertension or preeclampsia) seeks to evaluate a number of markers of maternal postpartum well-being, including maternal mood, breastfeeding, cognitive function, maternal-infant attachment, maternal perception of control, and postpartum pain between women who did and did not receive magnesium prophylaxis in the peripartum period.

This project will include 300 women recruited from the obstetrical service at Prentice Women's Hospital. Women will be included if they are at least 34 weeks gestation, have a singleton pregnancy, and have been diagnosed with a hypertensive disorder of pregnancy (either gestational hypertension or preeclampsia). Women will be exposed to magnesium for the indication of preeclampsia at the discretion of their obstetric provider.

Intrapartum baseline magnesium serum levels will be drawn for all women. For women who are receiving a magnesium infusion, serum magnesium levels will be repeated during the magnesium infusion (after receipt of the bolus infusion). For women who elect to receive neuraxial analgesia, CSF will be obtained and central magnesium levels drawn at the time of epidural placement.

Prior to discharge from the hospital, baseline demographic and clinical data will be obtained via chart review. Surveys will be administered to assess potential confounders of depression. A baseline self-reported depression survey, the Quick Inventory of Depressive Symptoms-Self Report (QIDS-SR) will be administered followed by a structured clinical interview for diagnosis (SCID), the gold standard for psychiatric research diagnosis. Women will be contacted at two weeks and again at six weeks postpartum and the QIDS-SR will be administered. For women with positive screens, a phone-based MINI will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant or immediately postpartum women
2. Age 18 and over
3. Singleton gestation
4. Diagnosis of hypertensive disorder of pregnancy
5. Gestational age of at least 34 weeks
6. English-speaking

Exclusion Criteria:

1. Women not meeting the above criteria
2. Prior receipt of magnesium during pregnancy
3. Intrauterine fetal demise or neonatal demise
4. Chronic hypertension

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This project will include 300 women recruited from the obstetrical service at Prentice Women's Hospital. Women will be included if they are at least 34 weeks gestation, have a singleton pregnancy, and have been diagnosis with a hypertensive disorder of pregnancy (either gestational hypertension or preeclampsia).
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Frequency of Postpartum Depression | Up to 6 weeks
  The frequency of postpartum depression at 2 weeks and 6 weeks postpartum

SECONDARY OUTCOMES:
Cognitive Function (measured using the Salthouse Digit Comparison and Size Judgment Span tests) | 4 days
  Immediate postpartum cognitive function
Pain (Self-reported) | 6 weeks
  Self-reported pain postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Emily S. Miller, MD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided